CLINICAL TRIAL: NCT06588582
Title: Exploring the Antecedents and Consequences of Cannabis Use in the Context of Coping: An Experimental Study
Brief Title: Perceptual Influences From Smoking Cannabis: an Experimental Study
Acronym: PISCES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carillon Skrzynski, Research Assistant Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-03-0215; 1K01DA058152-01A1 (NIH)
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Cannabis Use; Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold Water (Experimental)
  Interventions: Other: Water Temperature Variation - CW
- Warm Water (Placebo Comparator)
  Interventions: Other: Water Temperature Variation - WW

INTERVENTIONS:
Other: Water Temperature Variation - WW — Participants are assigned to warm water temperature.
  Arms: Warm Water
Other: Water Temperature Variation - CW — Participants are assigned to cold water temperature and are video recorded.
  Arms: Cold Water

SUMMARY:
The purpose of the study is to better understand the effects of cannabis in relation to mental and physical states including its relationship with mood, cognition, perception including the experience of temperature and pain, and heart rate.

We expect that participants will be in this research study for approximately one week. The total amount of time that participants will spend completing study tasks will be about 2.5 hours across two separate in-person visits.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age
* Endorsement of at least some use of cannabis for coping purposes (>1 on CMMQ)
* Regularly use flower cannabis products (i.e., ≥1x/week in the last 6 months)
* Proficient in English language
* At least occasional use of CBD+THC or CBD-dominant products (e.g., ≥1x/month)

Exclusion Criteria:

* Diagnosis or use of medications for substance use or psychotic disorders
* Report of other drug use (cocaine, opiates, methamphetamine) in the past 90 days or fail urine screen for any of these drugs
* Females cannot be pregnant or trying to become pregnant or nursing mothers
* Not able to provide informed consent

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Blood Cortisol Levels | Pre-Use/Pre-Water Task, 20 minutes Post-Use, 40 minutes Post-Use
  Cortisol levels are measured in blood.
Cannabis Used | Immediate Post-Use
  Grams of product used is calculated. Product is measured before and after use to measure how much was used.
Blood Endocannabinoid Levels | Pre-Use/Pre-Water Task, 20 minutes Post-Use
  Blood levels of AEA are measured.
Heart Rate | Pre-Use/Pre-Water Task, Pre-Use/Post-Water Task, 20 minutes Post-Use
  Participant HR is measured via pulse oximeter.
Social Anxiety | Pre-Use/Pre-Water Task
  Social Interaction Anxiety Scale (SIAS). 20 item survey, questions are answered on scale of 0 (not at all) to 4 (extremely), with higher scores indicating higher social anxiety. Questions are summed, with higher overall scores indicating higher social anxiety.
Inhibitory Control | Baseline
  Go/No-go Task. Participants are asked to complete a cognitive task where they see the text "Go" or "No go" during different trials. When they see "Go", they need to push a button within 2 seconds. When they see "No-go", they need to make sure they do not press the button (for 2 seconds). This is a measure of impulsivity.
Stress | Pre-Use/Pre-Water Task
  Stress Subscale of Depression and Anxiety Stress Scale measures stress. On scale from 0 (does not apply to me at all) to 3 (apply to me very much or most of the time). Higher scores indicate higher stress levels.
Blood cannabinoid levels | Pre-Use/Pre-Water Task, 20 minutes Post-Use
  THC and CBD blood levels are measured.
Current Pain | Pre-Use/Pre-Water Task, Pre-Use/Post-Water Task, 20 minutes Post-Use, 40 minutes Post-Use
  Internal scale/measure, measured from 0 (no pain) to 10 (worst pain imaginable). Participants report current pain on this self-report scale.
Mood | Pre-Use/Pre-Water Task, Pre-Use/Post-Water Task, 20 minutes Post-Use, 40 minutes Post-Use
  Profile of Mood States (POMS). Focus on the stress, anxiety, tension, and relaxation questions (combined for a tension/anxiety subscale). Questions are on a scale 1 (not at all) to 5 (extremely). Scores are summed, with higher scores indicating more tension/anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado at Boulder, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided